CLINICAL TRIAL: NCT03536832
Title: Comparison of Suture Materials for Subcuticular Skin Closure at Cesarean Delivery
Brief Title: Subcuticular Skin Closure at Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berna Aslan Cetin, Md, ObGYN, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018.4.20
Record Dates: First submitted 2018-05-09; First posted 2018-05-25 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-10

CONDITIONS: Cesarean Section; Infection
Keywords: Cesarean Section; Complications; suture material
MeSH Terms: conditions — Infections | interventions — Cesarean Section; Polyglactin 910

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cesarean section with Vicryl (Active Comparator): Women undergoing cesarean section with low transverse skin incisions will be closed with 3-0 Vicryl.
  Interventions: Procedure: Cesarean Section with Vicryl
- cesarean section with prolene (Active Comparator): Women undergoing cesarean section with low transverse skin incisions will be closed with 3-0 Prolen.
  Interventions: Procedure: Cesarean Section with Prolen

INTERVENTIONS:
Procedure: Cesarean Section with Vicryl — Pfnannenstiel incision will be done under general or spinal anaesthesia. The abdomen will be opened and fetus and plasenta will be delivered. Then abdomen will be closed. Skin will be closed with Vicryl.
  Arms: cesarean section with Vicryl
Procedure: Cesarean Section with Prolen — Pfnannenstiel incision will be done under general or spinal anaesthesia. The abdomen will be opened and fetus and plasenta will be delivered. Then abdomen will be closed. Skin will be closed with prolen.
  Arms: cesarean section with prolene

SUMMARY:
Subcuticular skin closure with suture after cesarean has been shown to result in lower rates of wound complications than with staple closure. However, the optimal choice of suture material for subcuticular skin closure is unclear. Vicryl vs Prolen suture materials will be used for subcuticular closure of transverse skin incisions after cesarean section. Patients will be controlled for superficial surgical site infections 1 week after the cesarean section.

DETAILED DESCRIPTION:
Cesarean section is the most common abdominal surgery worldwide. Subcuticular skin closure with suture after cesarean has been shown to result in lower rates of wound complications than with staple closure. However, the optimal choice of suture material for subcuticular skin closure is unclear. Vicryl vs Prolen suture materials will be used for subcuticular closure of transverse skin incisions after cesarean section. Patients will be controlled for superficial surgical site infections 1 week after the cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40
* women undergoing cesarean section

Exclusion Criteria:

* body mass index>30

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
surgical site infection | 1 week
  infection

CONTACTS AND LOCATIONS:
Overall Officials: Berna Aslan A Çetin, Principal Investigator — KSSTRH
Locations (1):
- Kanuni SSTRH, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided